CLINICAL TRIAL: NCT04832178
Title: Use of Sumor in the Antidepressant Therapy of Subjects With Major Depression: a Randomized Placebo-controlled Clinical Trial
Brief Title: Sumor as Adjuvant Therapy in Treatment-resistant Major Depression
Acronym: SUSCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Rotella, Dirigente Medico 1° livello - Psichiatra, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14976
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- SUMOR (Experimental)
  Interventions: Dietary Supplement: SUMOR

INTERVENTIONS:
Dietary Supplement: SUMOR — SUMOR is a food supplement distributed in Italy by ArcaPharma. regularly entered in the register of Food Supplements of the Ministry of Health (number 62590). Formulated in prolonged-release tablets, each tablet contains the following substances:
  * S-Adenosyl-L-Methionine sulfate p-toluenesulfonate 250 mg
  * Betaine hydrochloride 250 mg
  * Vitamin C 80 mg
  * Vitamin B1 1.1 mg
  * Vitamin B2 1.4 mg
  * Vitamin B6 1.4 mg
  * Vitamin B12 2,5 µg
  * Folic Acid 200 µg
  * Selenium 37 µg
  Arms: SUMOR
Other: Placebo — Placebo tablet will be identical in appearance to the experimental product (SUMOR).
  Arms: Placebo

SUMMARY:
Sumor is a food supplement that combines the main coenzymes of the S-Adenosyl methionine (SAMe) cycle, namely vitamins B6, B12 and folate, with SAMe and betaine. Sumor also contains vitamin C, a molecule that has shown promise in the treatment of depression in experimental models, and selenium, an antioxidant agent whose blood deficiency has been associated with depressive symptoms in some preliminary studies. There are no studies in the literature on the efficacy of this combination in the adjuvant therapy of depression. The purpose of this study is to compare the effects of Sumor in co-therapy with an SSRI antidepressant versus co-therapy with placebo in patients with treatment-resistant Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder according to DSM-5 criteria
* Treatment-resistant status, assessed by clinical interview, after four weeks after SSRI therapy prescription as per NICE guidelines (National Institute for Health and Care Excellence, 2009)
* Age between 18 and 65 years
* Signature of informed consent

Exclusion Criteria:

* Presence of intellectual disability or illiteracy
* Diagnosis of a disorder belonging to the spectrum of schizophrenia or other psychotic disorders according to DSM-5
* Diagnosis of a disorder belonging to the bipolar spectrum according to DSM-5
* Concomitant intake of therapy with other antidepressants, antipsychotics or mood stabilizers at the time of evaluation or in the previous 4 weeks
* State of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Baseline and 8 weeks
  The change in total HAM-D score between baseline and the 8-week follow-up was the primary outcomes measure. This measure is a clinician rated inventory of depressive symptoms. All items are scored on scales ranging from 0-2 to 0-4, and the sum of the scores provides the total score for the measure. On this scale, higher scores indicate poorer outcomes. Scores over 24 are considered indicative of severe depressive symptoms.

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Baseline, 2 weeks, and 4 weeks
  The change in total HAM-D score between baseline and the intermediate 2-week and 4-week follow-ups were considered secondary outcomes measures.
Hamilton Anxiety Scale (HAM-A) | Baseline, 2 weeks, 4 weeks and 8 weeks
  The change in total HAM-A score between baseline and the 2-week, 4-week and 8-week follow-ups were considered secondary outcomes measures. This measure is a clinician rated inventory of anxiety symptoms. The sum of the scores provides the total score for the measure. On this scale, higher scores indicate poorer outcomes.
SIDE | Baseline, 2 weeks, 4 weeks and 8 weeks
  A self-assessment questionnaire for undesirable effects in psychopharmacological treatment, developed by the Department of Psychiatry of Vanderbilt University in Nashville. It allows to investigate the presence or absence of 48 symptoms, exploring their severity and the relationship with the treatment.
Depressive symptoms remission | Baseline, 2 weeks, 4 weeks and 8 weeks
  Remission rate of Major Depression in the two groups over the course of treatment, defining remission as a score ≤ 7 on the HAM-D scale

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Rotella, PhD, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No